CLINICAL TRIAL: NCT05208827
Title: A Multicenter Randomized Controlled Study of Vitamin D Supplementation in Pregnant Women for the Prevention of Gestational Diabetes
Brief Title: Vitamin D Supplementation for the Prevention of GDM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GDM20211008
Record Dates: First submitted 2021-11-24; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Vitamin D; Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Randomized controlled study design
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Take two tablets once a day.Each tablet contains 800 units of vitamin D3, for a total of 1600 units taken orally daily
  Interventions: Drug: Vitamin D3
- Control Group (Placebo Comparator): The control group received the same packaged, similar-looking, similar-tasting placebo from the same manufacturer, containing starch, peanut oil (no pharmaceutical value)
  Interventions: Drug: The placebo(not contain vitamin D)

INTERVENTIONS:
Drug: Vitamin D3 — Participants began to take medication at 12 weeks of gestation, and participants in the second trimester began to take medication at the time point of enrollment.The dosage is 2 tablets per day, taken orally for 12 weeks.The drug in the intervention group was fat-soluble vitamin D3, which was produced by Sinopril Holding Starfish Pharmaceutical (Xiamen) Co., LTD. Each tablet contained 800 units of vitamin D3, vegetable oil and starch as auxiliary material.
  Arms: Experimental group
Drug: The placebo(not contain vitamin D) — Pills that looked, colored and tasted like vitamin D in the control group, but contained only starch and vegetable oil and no vitamin D.
  Arms: Control Group

SUMMARY:
This study was a double-blind multicenter randomized controlled study.

DETAILED DESCRIPTION:
This study intends to adopt a randomized controlled study design, and randomly divide pregnant women at high risk of GDM into intervention group (VitD3:1600 IU/ day) (n=800) and control group (placebo:2 tablets/day) (n=800) until the end of delivery. The risk of GDM in pregnant women of the two groups was compared, the preventive effect of high-dose VitD supplementation during pregnancy on different subtypes of GDM was determined, and the effects of VitD supplementation on VitD nutritional status during pregnancy and birth outcome and health of offspring were explored, so as to provide evidence-based basis for rational VitD supplementation during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are 8 to 14 weeks pregnant ; ② 18 to 45 years old; ③ Pregnant women at high risk of GDM (meeting any of the following conditions) : A) BMI ≥24 kg/m2 before or during pregnancy; B) family history of diabetes or GDM; C) Previous pregnancy diagnosed as GDM; D) with a history of macrosomia (≥4000 g); E) A history of abnormal glucose tolerance: 5.7-6.4% hBA1c or 6.1-7.0 mmol/L fasting blood glucose.

  * Sign informed consent. -

Exclusion Criteria:

* Patients with a history of diabetes or currently diagnosed diabetes (including type 1 and type 2 diabetes);

  * HBA1c ≥6.5% or fasting blood glucose & GT;7.0 mmol/L with obvious symptoms of diabetes;

    * Patients with current or past abnormalities in calcium metabolism (hypoparathyroidism/hyperthyroidism, kidney stones), high urinary calcium or hypercalcemia;

      * Daily VitD intake & GT;800 IU. ⑤ Suffering from serious chronic diseases (heart, lung, liver, kidney and other dysfunction) or mental illness;

        * They cannot walk 100 meters safely; 7. Multiple pregnancies or assisted reproduction; ⑧ need complex diet;

          * Cannot speak Mandarin fluently; ⑩ Those who are participating in other clinical trials or who are considered unsuitable for clinical trials by researchers for other reasons.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study only applied to women with normal pregnancies
Enrollment: 1600 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes | At 24-28 weeks of gestation
  We will judge whether patients have gestational diabetes based on OGTT results (fasting, 1-hour, 2-hour blood glucose results) .

SECONDARY OUTCOMES:
Newborn birth weight | immediately after delivery
  Weight of newborn at birth
Gestational age | immediately after delivery
  Determine the gestational age of the woman and whether preterm birth exists
Weight gain during pregnancy | First day after birth
  Weigh the pregnant woman on the first day after delivery and subtract her weight before pregnancy from the birth examination book

CONTACTS AND LOCATIONS:
Overall Officials: Danqing Chen, doctor, Study Chair — Obstetrics and Gynecology Hospital affiliated to Zhejiang University School of Medicine
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China